CLINICAL TRIAL: NCT04804397
Title: Effects of Sucrose Added Blind to the Diet Over Eight Weeks on Body Mass and Weight in Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Responsible Party: Principal Investigator, Richard Hammersley, Professor of Health Psychology, University of Hull
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PSY4272
Record Dates: First submitted 2016-01-26; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Overweight
Keywords: Sucrose; Sugar; Carbohydrate; Weight gain; men
MeSH Terms: conditions — Overweight; Weight Gain; Multiple Endocrine Neoplasia Type 1 | interventions — Sucrose; Aspartame

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sucrose (Experimental): Sucrose: 1l sucrose sweetened soft drink per day for 8 weeks (1650 KJ, 97g carbohydrate per day) as 4 25cl drinks
  Interventions: Dietary Supplement: Sucrose
- Aspartame (Placebo Comparator): Aspartame: 1l aspartame sweetened soft drink per day for 8 weeks as 4 25cl drinks
  Interventions: Dietary Supplement: Sucrose

INTERVENTIONS:
Dietary Supplement: Sucrose — Sucrose sweetened soft drinks
  Other Names: Aspartame; Aspartame sweetened soft drinks as comparator

SUMMARY:
Background: Sugar intake, especially in liquid, correlates with obesity. Yet, whether it is a special cause of obesity is less clear. Few experimental studies exist.

Aim: To replicate the investigators' previous 4 week experiments on women with men over 8 weeks to ascertain if: they gain weight given sucrose soft drinks; mood is affected; energy intake is affected.

Participants: 80 men BMI 25-35, aged 30-55. Procedure: After a week of baseline, over eight weeks single blind 40 men received soft drinks containing sucrose (1650 KJ, 97g carbohydrate per day), 40 received control drinks. A three-day food diary with mood ratings and activity levels was completed during baseline and weeks 1, 4 and 8 of the experiment. Body mass was recorded weekly with other anthropometric measures.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-35

Exclusion Criteria:

* Diabetes,
* other health problems,
* medication,
* dislike of soft drinks

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Body Mass | Eight Weeks
  Do participants gain weight?

SECONDARY OUTCOMES:
Daily energy intake assessed by free-living unweighed food diary | Eight Weeks
  Do participants eat less to compensate for added sucrose?
Mood assessed using 10 rating scales | Eight Weeks
  Are there changes in rated mood during sucrose supplementation?

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hammersley, PhD, Study Chair — University of Hull

IPD SHARING:
Plan to Share IPD: No